CLINICAL TRIAL: NCT05030376
Title: Comparative Effects of Intraileal Glucose vs. Saline Infusion on Hormone Secretion and Glycemic Excursions in Subjects With Ileostomy
Brief Title: Intraileal Glucose vs. Saline Infusion on Hormone Secretion and Glycemic Excursions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong First Medical University (Other)
Responsible Party: Principal Investigator, Sanyuan Hu, Professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: QLYY-CRC-2020-001
Record Dates: First submitted 2021-08-23; First posted 2021-09-01 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Incretins

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with ileostomy without type 2 diabetes (Experimental): intraileal glucose or saline infusion via ileostomy
  Interventions: Dietary Supplement: intraileal infusion
- patients with ileostomy with type 2 diabetes (Experimental): intraileal glucose or saline infusion via ileostomy
  Interventions: Dietary Supplement: intraileal infusion

INTERVENTIONS:
Dietary Supplement: intraileal infusion — intraileal glucose or intraileal saline infusion

SUMMARY:
The distal ileum, where the glucagon-like peptide 1 (GLP-1) releasing cells predominate, is an important organ in mediating glycemic control. However, the distal ileum is not easy to access and the correspond in vivo research remains to be difficult. The investigators intend to recruit subjects who underwent rectal surgery with simultaneous protective ileostomy and evaluate hormone secretion and glycemic excursions via ileostomy glucose or saline infusion, and quantify the glucose absorption rate within the distal ileum.

ELIGIBILITY:
Inclusion Criteria:

* Male and postmenopausal females aged 18 - 75 years
* Body mass index (BMI) 20 - 35 kg/m2
* With protective ileostomy due to benign or malignant rectal surgery

Exclusion Criteria:

* History of postoperative adjuvant chemotherapy
* Other significant illness, including epilepsy, cardiovascular or respiratory disease
* Impaired renal or liver function (as assessed by calculated creatinine clearance < 90 mL/min or abnormal liver function tests (> 2 times upper limit of normal range))
* Donation of blood within the previous 3 months
* Participation in any other research studies within the previous 3 months
* Females who are pre-menopausal
* Inability to give informed consent
* Vegetarians

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
serum or plasma GLP-1 changes during intraileal infusion | 180 minutes
  concentration of serum or plasma GLP-1 (pmol/L)
serum or plasma GIP changes during intraileal infusion | 180 minutes
  concentration of serum or plasma GIP (pmol/L)
serum or plasma ghrelin changes during intraileal infusion | 180 minutes
  concentration of serum or plasma ghrelin (pg/ml)
serum or plasma c-peptide changes during intraileal infusion | 180 minutes
  concentration of serum or plasma c-peptide (pmol/L)
serum or plasma insulin changes during intraileal infusion | 180 minutes
  concentration of serum or plasma insulin (pmol/L)
serum or plasma glucagon changes during intraileal infusion | 180 minutes
  concentration of serum or plasma glucagon (pmol/L)
glucose absorption capacity | 180 minutes
  estimated glucose absorption rate during intraileal glucose infusion

CONTACTS AND LOCATIONS:
Overall Officials: Kexin Wang, Study Director — Qilu Hospital of Shandong University
Locations (2):
- China (2):
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - the first affiliated hospital of Shandong First Medical University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang X, Cheng Z, Dong S, Rayner C, Wu T, Zhong M, Zhang G, Wang K, Hu S. Effects of ileal glucose infusion on enteropancreatic hormone secretion in humans: relationship to glucose absorption. Metabolism. 2022 Jun;131:155198. doi: 10.1016/j.metabol.2022.155198. Epub 2022 Apr 6. PMID 35395220